CLINICAL TRIAL: NCT00639054
Title: The Molecular Characterization of Multiple Myeloma at Relapse
Acronym: MM-FISH/DNA
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Herlev Hospital (Other); Zealand University Hospital (Other); Naestved Hospital (Other); Agnes og Poul Friis Fond (Unknown); Carl og Ellen Hertzs Legat til Dansk Læge- og Naturvidenskab (Unknown); Dagmar Marshalls Fond (Unknown); Danish Cancer Research Foundation (Other); Direktør Jacob Madsen og hustru Olga Madsens Fond (Unknown); Elna og Jørgen Fagerholt Pedersens Kræftforskningsfond (Unknown); Eva og Henry Frænkels Mindefond (Other); Manufacturer Einar Willumsen's memorial team (Other); Fonden til Lægevidenskabens Fremme (Other); Grosserer M. Brogaard og Hustrus Mindefond (Unknown); Højmosegård-Legatet (Unknown); Janssen-Cilag, S.A. (Industry); Karen A. Tolstrups fond (Unknown); Krista og Viggo Petersens Fond (Unknown); Købmand Sven Hansen og hustru Ina Hansens Fond (Unknown); Meta og Håkon Baggers Fond (Unknown); Reinholdt W. Jorck og hustrus Fond (Unknown)
Responsible Party: Principal Investigator, N. Emil U. Hermansen, Ph.D student, Rigshospitalet, Denmark
Other Study IDs: 959593931/Emil Hermansen; H-B-2007-117 (Other: The National Committee on Health Research Ethics (Denmark))
Record Dates: First submitted 2008-03-11; First posted 2008-03-19 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Multiple Myeloma
Keywords: classification; diagnosis; genetics; mortality; pathology
MeSH Terms: conditions — Multiple Myeloma; Disease | interventions — Bone Marrow Examination; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral whole blood Bone marrow
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Newly diagnosed patients: Newly diagnosed high-dose therapy candidates. Participation means bone marrow examination (donating 7.5 ml of fresh bone marrow) and blood samples (24 ml of peripheral blood) for biochemical and genetic analyses regarding multiple myeloma, and granting access to clinical data relating to multiple myeloma.
  Interventions: Procedure: Bone marrow examination; Procedure: Blood samples
- Relapse patients: Formerly high-dose treated patients with progressive disease. Participation means bone marrow examination (donating 7.5 ml of fresh bone marrow) and blood samples (24 ml of peripheral blood) for biochemical and genetic analyses regarding multiple myeloma, and granting access to clinical data relating to multiple myeloma.
  Interventions: Procedure: Bone marrow examination; Procedure: Blood samples
- Healthy controls: Healthy blood and bone marrow donors. Participation means bone marrow examination (donating 7.5 ml of fresh bone marrow) for genetic analyses serving to compare normal bone marrow with bone marrow from multiple myeloma patients.
  Interventions: Procedure: Bone marrow examination

INTERVENTIONS:
Procedure: Bone marrow examination — 7.5 ml of iliac crest bone marrow drawn in addition to diagnostic samples.
Procedure: Blood samples — 24 ml of cubital vein blood drawn in addition to diagnostic samples.
  Groups: Newly diagnosed patients; Relapse patients

SUMMARY:
Observational study investigating prognostic factors in newly diagnosed and relapsed multiple myeloma patients by use of clinical data, biochemical markers (blood samples), cytogenetic markers and gene expression profiling (myeloma cells from fresh bone marrow samples). Enabling future genetic studies by establishing a biobank of bone marrow and peripheral blood samples.

DETAILED DESCRIPTION:
Multiple myeloma (MM) is an incurable cancer. The disease can often be brought to a halt with chemotherapy which in younger patients is accompanied by stem cell transplantation. But the disease relapses almost invariably. Cytogenetic changes in the myeloma cells can serve as prognostic markers. Accordingly, 25% of the patients show changes associated with a prognosis so poor that they should probably receive experimental treatment right from the start. Nevertheless, a part of these patients survive much longer than expected. Thus, the prognosis must depend on additional genetic events.

The aim of this project is to widen the investigators knowledge of the nature, chronology and prognostic value of the genetic events in MM in order to improve the risk stratification of the patients and hence the choice of treatment. Using cytogenetics (interphase FISH) and molecular biological analyses (SNP, GEP, miRNA) the investigators will study the changes in the myeloma cells. The investigators will search for genetic and clinical differences between patients within the same cytogenetic group and between patients at diagnosis and at relapse. The study population will consist of 100 newly diagnosed patients and 100 relapse patients included prospectively over a 2-year period in a cooperation between the four departments of hematology in Zealand, Denmark.

Hypotheses:

1. Early relapse depends on a) molecular defects in the myeloma cells detectable with FISH, GEP, SNP and/or miRNA analyses, and b) the acquisition of new mutations resulting in chemotherapy resistance and increased prolific capacity.
2. The progressive reduction of event free survival seen with every relapse until the disease turns refractory can be explained by selection of critical mutations.
3. The cytogenetic changes associated with poor prognosis represent a heterogenous group of patients in whom the responsible genetic events remain unknown.

ELIGIBILITY:
Inclusion Criteria:

* patients newly diagnosed with multiple myeloma and at the same time eligible for high dose chemotherapy and autologous stem cell transplantation
* patients with multiple myeloma experiencing relapse after high dose chemotherapy and autologous stem cell transplantation

Exclusion Criteria:

* for newly diagnosed patients: age or comorbidity preventing high dose chemotherapy and autologous stem cell transplantation,
* for all patients: age below 18, physical or psychological incapability to give an informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed and/or treated at departments of hematology. Healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2008-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Molecular characteristics (by FISH, SNP, GEP, miRNA) | 0-3 years

SECONDARY OUTCOMES:
Event free survival (EFS) | 0-10 years
Overall survival (OS) | 0-10 years

CONTACTS AND LOCATIONS:
Overall Officials: N Emil U Hermansen, MD, Principal Investigator — Rigshospitalet, Denmark; Peter Gimsing, MD, DMSc, Study Chair — Rigshospitalet, Denmark; Annette J Vangsted, MD, DMSc, Study Chair — Zealand University Hospital; Mette K Andersen, MD, DMSc, Study Chair — Rigshospitalet, Denmark; Finn C Nielsen, MD, DMSc, Study Chair — Rigshospitalet, Denmark; Dan Kristensen, MD, Study Chair — Naestved Hospital, Denmark; Nielsaage T Clausen, MD, Study Chair — Herlev Hospital
Locations (1):
- Multiple Myeloma Research Laboratory, Dept Hematology, Cph Univ Hosp Rigshospitalet, Copenhagen, Capital Region, Denmark

REFERENCES:
- [Derived] Hermansen NE, Borup R, Andersen MK, Vangsted AJ, Clausen NT, Kristensen DL, Nielsen FC, Gimsing P. Gene expression risk signatures maintain prognostic power in multiple myeloma despite microarray probe set translation. Int J Lab Hematol. 2016 Jun;38(3):298-307. doi: 10.1111/ijlh.12486. Epub 2016 Mar 29. PMID 27027250